CLINICAL TRIAL: NCT04894513
Title: Electro Physiological Responses to Kabat Motor Control Re-education on Bell's Palsy: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lama Saad El-Din Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T./REC /012/003143
Record Dates: First submitted 2021-04-13; First posted 2021-05-20 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Facial Nerve Palsy; Bell's Palsy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Intervention Model Description: control group which received conventional selected program, and study group received the same exercise training program in addition to Kabat motor control re-education therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the study group received the conventional selected program in addition to Kabat motor control re-education
  Interventions: Other: Kabat motor control re-education therapy; Other: conventional selected program
- control group (Experimental): the control group received the conventional selected program
  Interventions: Other: conventional selected program

INTERVENTIONS:
Other: Kabat motor control re-education therapy — Kabat motor control re-education therapy that includes specific movements with predefined patterns of facial muscles exercises, which is spiral and diagonal movements involve the facial muscles, which are brought to train in global patterns. The program of treatment for three times per week for six weeks.
  Arms: study group
Other: conventional selected program — the conventional selected program in the form of electrical stimulation (Faradic current) of affected muscles, facial muscle exercise program in front of the mirror, and home advices.

SUMMARY:
To investigate the Effect of Kabat motor control re-education therapy on facial nerve Electro physiological responses and facial muscles function in bell's palsy.

BACKGROUND: facial nerve recovery in children could be improved through facilitation of nerve regeneration which can be enhanced through Kabat motor control re-education therapy.

DETAILED DESCRIPTION:
Thirty children with bell's palsy will participate in this study. The patients will randomly be divided into two equal groups; the control group received the conventional selected program, and the study group received the same exercise training program in addition to Kabat motor control re-education therapy. The program of treatment will be three times per week for six weeks.

The evaluation methods: Facial nerve distal latency, amplitude, and percentage of degenerations via the Neuropack S1 MEB9004 EMG device, the Facial Disability Index, and Sunnybrook facial grading system (SBFGS) all the assessment methods before the program and after finishing the program

ELIGIBILITY:
Inclusion Criteria:

* Thirty child diagnosed as acquired bell's palsy with unilateral peripheral facial paralysis
* Both gender
* Their age ranged from 12:16 years old.

Exclusion Criteria:

* difficulty to communicate or to understand program instructions
* Oral dentures, Skin infection and metal implants on face
* Sensory loss over the face, Recurrent facial paralysis
* any other disorders or neurological deficits,
* a history of surgical intervention for the ear and facial nerve palsy
* pain of any other origin
* non co-operative patients

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Electroneurography | 6 weeks
  Measuringthe Facial nerve distal latency measured in millisecond (ms).via the Neuropack S1 MEB9004 EMG device
Electroneurography | 6 weeks
  Measuring the Facial nerve amplitude measured in (mv).via the Neuropack S1 MEB9004 EMG device
Electroneurography | 6 weeks
  Measuring the Facial nerve percentage of degenerations measured in(%).via the Neuropack S1 MEB9004 EMG device

SECONDARY OUTCOMES:
Sunnybrook facial grading system (SBFGS) | 6 weeks
  it is a clinical grading system of facial function in facial palsy. It consists of 13 items-3 resting, 5 voluntary movement and 5 synkinesis items-answered on categorical answering scales. A SB composite score (range 0-100) and resting symmetry (range 0-20), voluntary movement (range 20-100) and synkinesis subscores (0-15) can be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamed SA, Saad El-Din Mahmoud L, Magdy ElMeligie M, Zoheiry IM. Electrophysiological responses to Kabat motor control re-education on Bell's Palsy: A randomized controlled study. J Musculoskelet Neuronal Interact. 2023 Mar 1;23(1):90-97. PMID 36856104